CLINICAL TRIAL: NCT04727177
Title: Precision-targeted Transcranial Magnetic Stimulation in the Treatment of Primary Dystonia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Hangzhou Normal University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SAHZhejiangU2
Record Dates: First submitted 2021-01-24; First posted 2021-01-27 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-01

CONDITIONS: Primary Dystonia; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Dystonic Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Transcranial magnetic stimulation — Transcranial magnetic stimulation (TMS) is a noninvasive biological stimulation technique born in the middle of 1980's.

SUMMARY:
In this scheme, TMS treatment of Primary dystonia is planned by precise magnetic resonance positioning.

ELIGIBILITY:
Inclusion Criteria:

* Primary dystonia

Exclusion Criteria:

* None

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Burke-Fahn-Marsden dystonia rating scale | Five days
  The BFMMS measures dystonia in nine body regions (including the eyes, mouth, speech and swallowing, neck, trunk, arms, and legs) with scores ranging from 0 (minimum) to 120 (maximum).The higher scores mean a worse outcome.
  The BFMDS is a functional marker consisting of parental- or self-reported daily activities (involving speech, handwriting,feeding, eating, swallowing, hygiene, dressing, and walking),with scores ranging from 0 (completely independent) to 30 (completely dependent).

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Feng, Principal Investigator — Zhejiang University
Locations (1):
- Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No